CLINICAL TRIAL: NCT05145075
Title: Surveying the Receptivity for Telemedicine Pre-operative Consultation in UZ Brussel.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Tele Pre-op Consultation
Record Dates: First submitted 2021-12-02; First posted 2021-12-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Remote Consultation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survey group (Experimental): Patients are asked to fill in a survey.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Patients are asked to fill in a survey concerning teleconsultations

SUMMARY:
We will be surveying patients coming to UZ Brussels for their pre-operative consultation, how they feel about changing these consultations to teleconsultations.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to a planned in-hospital pre-operative consultation at UZ Brussels.

Exclusion Criteria:

* Language barrier
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Willingness to have a teleconsultation: Survey | 4 months
  Would this person be willing to have a teleconsultation in stead of a consultation face to face

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided